CLINICAL TRIAL: NCT03980548
Title: Targeting Mitochondrial Fusion and Fission to Prevent Atherosclerosis: Getting the Balance Right - MITOFFA
Brief Title: Targeting Mitochondrial Fusion and Fission to Prevent Atherosclerosis: Getting the Balance Right
Acronym: MITOFFA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/2497; SHF/FG651P/2017 (Other Grant/Funding Number: SingHealth Foundation)
Record Dates: First submitted 2019-06-06; First posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2018-08

CONDITIONS: CAD Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Tissue samples: LIMA or radial or aorta or aortic valve
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- CABG patients
  Interventions: Procedure: CABG
- PAD patients
  Interventions: Procedure: CABG
- Healthy volunteers
  Interventions: Procedure: CABG
- Patients with CAD
  Interventions: Procedure: CABG

INTERVENTIONS:
Procedure: CABG — Patients undergoing coronary artery bypass graft and patient presented with ACS undergoing PCI
  Other Names: PCI

SUMMARY:
Our preliminary data suggests that pharmacological inhibition of the mitochondrial fission protein, Drp1, reduced atherosclerotic plaque volume and attenuated macrophage accumulation within the plaque in an ApoE-/- mouse model of wire-induced carotid arterial injury. Furthermore, we hypothesize that modulation of mitochondrial morphology and metabolism with Drp1 inhibition prevents atherosclerosis by reducing monocyte activation and migration. In this research proposal, our overall objective will be to investigate the role of Drp1 in human monocytes and macrophages as novel therapeutic targets for preventing atherosclerosis.

DETAILED DESCRIPTION:
Study 1 (tissue sample study): To investigate the changes in mitochondrial function and pro-inflammatory markers in human arterial atherosclerotic plaques.

Hypothesis: Macrophages from femoral artery atherosclerotic plaques in patients with peripheral artery disease will display upregulation of mitochondrial fission proteins and features of pro-inflammatory activation.

Study 2 (white blood cell study): To investigate the changes in mitochondrial function and pro-inflammatory markers in white blood cells from patients with stable and unstable coronary artery didease (CAD).

Hypothesis: Monocytes from patients with unstable CAD will display upregulation of Drp1 and features of pro-inflammatory activation, mitochondrial fission, impaired mitochondrial respiratory function, and perturbed metabolism, when compared to monocytes from patients with stable CAD.

ELIGIBILITY:
Inclusion Criteria:

Study 1 (tissue sample study):

CABG patients

1. Patients aged ≥21 years old
2. Undergoing elective CABG with aortic valve surgery

PAD patients:

1. Patients aged ≥21 years old
2. Undergoing either elective surgical femoral or carotid endarterectomy

Study 2 (white blood cell study):

1) Healthy volunteers aged ≥21 years old 2) Patients with stable CAD 3) Patients admitted with ACS treated by PCI in prior 24 hours.

-

Exclusion Criteria:

1. General exclusion criteria will be a known history of leucopenia, thrombocytopenia, or severe hepatic or renal dysfunction, as well as evidence for inflammatory or malignant disease.
2. History of haematological disorders
3. Cardiac arrest, Cardiogenic shock, Poor pre-morbid status, Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study 1 (tissue sample study):
  * 25 adult patients undergoing coronary artery bypass graft (CABG) surgery: Control tissue will be collected from the left internal mammary artery (LIMA) or radial artery (RA) Atherosclerotic tissue will be collected from aortic root
  * 25 adult patients undergoing surgical femoral or carotid endarterectomy Endarterectomy atherosclerotic tissue will be collected
  Study 2 (white blood cell study):
  * 50 healthy adult volunteers Control blood sample will be collected
  * 50 adult patients with stable CAD Stable CAD blood sample will be collected
  * 50 adult patients with unstable CAD Unstable CAD blood sample will be collected
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
"mitochondria-shaping" proteins expression quantified on immunoblotting in patients with atherosclerosis disease. | 2 years
  Primary outcome analysis for aim 1:
  The primary endpoint is "mitochondria-shaping" proteins expression quantified on immunoblotting in patients with atherosclerosis disease. The statistical analysis will be performed by 2-tailed student's T-test with the platelet "mitochondria-shaping" proteins expression as the response variable. The primary analyses will be by per protocol analysis and there will also be an intention to treat analysis.
  Primary outcome analysis for aim 1:
  The primary endpoint is "mitochondria-shaping" proteins expression quantified on immunoblotting in patients with atherosclerosis disease. The statistical analysis will be performed by 2-tailed student's T-test with the platelet "mitochondria-shaping" proteins expression as the response variable. The primary analyses will be by per protocol analysis and there will also be an intention to treat analysis.
  The primary endpoint is "mitochondria-shaping" proteins expression quantified on immunoblotting in patients

CONTACTS AND LOCATIONS:
Locations (1):
- Hector A. Cabrera-Fuentes, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided